CLINICAL TRIAL: NCT00938886
Title: Naltrexone for At-Risk and Problem Drinking in Smoking Cessation Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Christopher W. Kahler, Professor of Behavioral and Social Sciences, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAA-17181-1
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Hazardous Drinking; Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Experimental): 50 mg daily naltrexone for 10 weeks
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Daily matched placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Daily 50 mg naltrexone
  Arms: Naltrexone
Drug: Placebo — Matched naltrexone placebo
  Arms: Placebo

SUMMARY:
To test whether naltrexone compared to placebo can reduce heavy drinking and improve smoking cessation outcomes in heavy drinkers seeking smoking cessation treatment.

DETAILED DESCRIPTION:
A substantial portion of individuals seeking behavioral and pharmacological treatment for smoking cessation drink excessively with many reporting significant alcohol problems. Although these at-risk and problem drinkers are unlikely to choose abstinence from alcohol as a goal, many make substantial reductions in their drinking during and after their quit smoking attempt. Thus, the context of smoking cessation treatment offers a unique and valuable opportunity in which to apply brief interventions and pharmacotherapy to catalyze change in excessive drinking in a population with markedly elevated risk for negative health outcomes. In our recent randomized clinical trial, standard smoking cessation treatment that incorporated a brief alcohol intervention showed promise in reducing drinking as well as in improving smoking cessation outcomes among heavy drinkers. However, these effects were relatively modest, especially among the heaviest drinkers, indicating that further study is warranted of methods to address heavy drinking in smoking cessation including the use of relevant pharmacotherapy. Naltrexone, in particular, shows promise for this purpose.

The overall aim of this project is to test the efficacy of naltrexone as a pharmacotherapy for excessive drinking when delivered to at-risk or problem drinkers who are seeking smoking cessation treatment. The proposed clinical trial uses a between-subjects design in which 300 at-risk or problem drinkers seeking treatment for smoking cessation will be randomly assigned to receive either daily 50 mg naltrexone or placebo. Medication will be initiated 2 weeks prior to participants' smoking quit date and continue for 10 weeks. All participants also will receive transdermal nicotine patch and a counseling and medication management intervention that provides advice for smoking cessation, advice regarding the effects of heavy drinking on both smoking cessation and health, and monitoring and encouragement of compliance with medications. Drinking and smoking outcomes will be assessed at 2, 8, 16, and 26 weeks after participants' smoking quit date. The primary aim of the study is to test the hypothesis that naltrexone will result in greater reductions in heavy drinking relative to placebo. The secondary aim will test whether naltrexone results in superior smoking outcomes relative to placebo, and tertiary aims will examine interrelationships among motivation for changing drinking, compliance with naltrexone, and drinking and smoking outcomes.

This study represents the first of its kind to provide naltrexone in conjunction with an opportunistic brief alcohol intervention for at-risk and problem drinkers not seeking alcohol treatment. Testing the potential benefits of naltrexone among at-risk and problem drinkers who smoke is of very high significance for public health efforts to reduce the markedly elevated rates of morbidity and mortality observed in this large, yet relatively understudied group.

ELIGIBILITY:
Inclusion Criteria:

* 1.) be at least 18 years of age, 2.) drink heavily at least once per month on average (≥4 drinks per occasion for women; ≥5 drinks for men), 3.) have smoked cigarettes regularly for at least one year, 4.) currently smoke at least 5 cigarettes a day, 5.) currently be using no other tobacco products or nicotine replacement therapy

Exclusion Criteria:

* 1.) meet criteria for current substance dependence (excluding nicotine and alcohol); 2.) report opiate use in the past month, have a drug screen positive for opiates, or require opiate containing medications for pain management; 3.) meet criteria for a current major depressive or manic episode; 4.) are currently psychotic or suicidal; 5.) have an unstable or serious medical condition that would preclude use of the nicotine patch or naltrexone (e.g., unstable angina pectoris, severe arrhythmia, recent congestive heart failure); 6.) have aspartate aminotransferase or alanine aminotransferase levels of more than 3 times the reference range or elevated bilirubin levels; or 7.) are currently pregnant or lactating, intend to become pregnant, or are not using a reliable means of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. Kahler, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Providence, RI and the surrounding community through bulletin board, radio, internet, newspaper, and public transportation advertisements.
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 75 | 75
Attended 1 Counseling Session | 70 | 70
Completed | 68 | 65
Not Completed | 7 | 10
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.7) | 41.8 (12.9) | 42.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 29 | 62
  Male | 42 | 46 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 73 | 67 | 140
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 12 | 25
  White | 55 | 54 | 109
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 1 | 2 | 3
Current Alcohol Dependence [Count of Participants; unit: Participants] | 23 | 19 | 42
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 0 to 10 where higher values indicates higher levels of nicotine dependence.
  units on a scale | 5.3 (2.2) | 5.4 (2.3) | 5.3 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days
Description: Defined for women as percent of days drinking 4 or more drinks in a day. For men, percent of days drinking 5 or more drinks in a day
Time Frame: Across the 6 months following smoking quit date
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 68 | 65
percentage of days | 11.1 (13.1) | 11.4 (11.3)

2. Secondary Outcome: 7-day Point Prevalence Smoking Abstinence
Description: Self-report abstinence from smoking over the past 7 days biochemically confirmed with carbon monoxide and saliva cotinine.
Time Frame: 26 weeks after target quit smoking date
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 75 | 75
Participants | 9 | 9

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 1/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 2/75
Other Adverse Events (participants affected / at risk) | 30/75 | 36/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=75) | Placebo (N=75)
Appendectomy (General disorders) | 0 (0) | 1 (1) — Emergency appendectomy
Back Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Back surgery to relieve acute nerve problem
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=75) | Placebo (N=75)
Nausea (Gastrointestinal disorders) | 8 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7) | 7 (7)
Adbominal pain (Gastrointestinal disorders) | 5 (5) | 7 (7)
Decreased appetite (Gastrointestinal disorders) | 5 (5) | 3 (3)
Headache (General disorders) | 4 (4) | 10 (10)
Dizziness (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 5 (5) | 7 (7)
Anxiety (Psychiatric disorders) | 8 (8) | 11 (11)
Insomnia (General disorders) | 11 (11) | 19 (19)
Somnolence (General disorders) | 9 (9) | 16 (16)
Depression (Psychiatric disorders) | 9 (9) | 7 (7)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes